CLINICAL TRIAL: NCT01796041
Title: A Phase 0/1, Open-Label, Single Center Study of the Imaging Potential of Indocyanine Green in Subject Undergoing Breast Cancer Surgery
Brief Title: Intraoperative Imaging of Breast Cancer With Indocyanine Green
Acronym: ICG
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 12111; 813695 (Other: UPenn IRB Protocol #)
Record Dates: First submitted 2013-01-18; First posted 2013-02-21 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2018-02

CONDITIONS: Invasive Ductal Carcinoma; Invasive Lobular Carcinoma; Ductal Carcinoma
MeSH Terms: conditions — Carcinoma, Lobular; Carcinoma, Ductal | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV Injection of ICG (Experimental)
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green
  Other Names: ICG; The chemical formula is C45H47N2O6S2Na

SUMMARY:
According to the World Health Organization, breast cancer is the most common cancer in women, and is responsible for 686,000 new cases every year. The WHO also posit that nearly 420,000 women perished from the disease in 2002. Surgery remains the best option for patients presenting with operable Stage I, II or III cancers. Breast conservation surgery has been shown to be as efficacious as mastectomy. About 60-70% of these women with operable breast cancer are breast conservation candidates. However, the need to achieve negative tumor margins often requires a second operation (re-excision) in up to 70% of the women having lumpectomy surgery. Currently, tumor margins assessment in the operating room is often assessed grossly by palpation. The ability to evaluate tumor margin using our proposed intraoperative imaging technique may provide the surgeon with an alternative, and hopefully, more sensitive method to assess tumor margins which may decrease re-excision and the morbidity associated with additional surgery, and, perhaps, lower the risk of local regional recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over 18 years of age
2. Women with newly diagnosed, operable invasive ductal carcinoma, invasive lobular carcinoma or ductal carcinoma who are deemed breast conservation surgery candidates (i.e. lumpectomy +/- sentinel node biopsy).
3. Breast cancer needs to be unifocal as determined by clinical parameters, e.g. by palpation or by breast imaging findings including mammogram, US and/or breast MRI. Multifocal disease, i.e. cancer confined to one quadrant, is eligible if patients are deemed breast conservation candidates.
4. Subject capable of giving informed consent and participating in the process of consent.

Exclusion Criteria:

1. Newly diagnosed breast cancer patients who are not breast conservation candidates and those with multicentric breast cancer (breast cancer documented in multiple quadrants by breast imaging or exam)
2. Pregnant women as determined by urinary or serum beta human chorionic gonadotropin (hCG) within 72 hours of surgery
3. Subjects with a history of iodide allergies
4. At-risk patient populations

   1. Homeless patients
   2. Patients with drug or alcohol dependence
   3. Patients unable to participate in the consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-07; Primary Completion 2016-11-09 (Actual); Study Completion 2016-11-09 (Actual)

PRIMARY OUTCOMES:
Identification | After infusion of ICG
  The primary outcome will be the proportion of patient's tumors identified by ICG uptake versus the proportion of patients identified by visual and tactile methods by the surgeon (considered standard of care)

SECONDARY OUTCOMES:
Evaluation | 0-5 years after surgery
  a) Correlate detected ICG excitation in shave lumpectomy margins with quantity of residual disease in histologic sections.
Evaluation | 0-5 years after surgery
  b) evaluate the rate of re-excision in participants compared to a matched case- control cohort with similar clinicopathological characteristics undergoing breast conservation surgery.
Evaluation | 0-5 years after surgery
  C) evaluate progression free survival in our study cohorts

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States